CLINICAL TRIAL: NCT06020651
Title: Vascular Toxicities of Immune ChecKpoint Inhibitors : From Bed to Benchside
Acronym: VICKI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CARDIO 05 2022
Record Dates: First submitted 2023-07-27; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-07

CONDITIONS: Renal Cell Carcinoma; Bladder Cancer; MSI-H Cancer; Cancer
Keywords: Atherosclerosis; Cancer; Immune Checkpoint Inhibitor; Vascular Diseases
MeSH Terms: conditions — Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Neoplasms; Atherosclerosis; Vascular Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: All participants will undergo the same cardiovascular assessment; only cancer therapies differ according to standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ICIs alone (Experimental): Participants on ICIs alone
  Interventions: Diagnostic Test: Arterial Doppler for Flow Mediated Reserve measurement
- ICIs + VEGF inhibitors (Experimental): Participants on ICIs + VEGF inhibitors
  Interventions: Diagnostic Test: Arterial Doppler for Flow Mediated Reserve measurement
- ICIs + chemotherapy (Experimental): Participants on ICIs + chemotherapy
  Interventions: Diagnostic Test: Arterial Doppler for Flow Mediated Reserve measurement
- Controls (Sham Comparator): Participants on other than ICIs cancer therapies
  Interventions: Diagnostic Test: Arterial Doppler for Flow Mediated Reserve measurement

INTERVENTIONS:
Diagnostic Test: Arterial Doppler for Flow Mediated Reserve measurement — Arterial Doppler (ultrasound, no radiation, no contrast agent) and blood sampling twice for participants on ICIs
  Other Names: Blood sampling

SUMMARY:
Immune checkpoint inhibitors (ICIs) are largely prescribed in a growing number of cancer diseases and at earlier stages (non metastatic cancer). Among immune-related adverse events, (iRAEs), the incidence of major cardiovascular events due to atherosclerosis reaches 13% at one year in patients at high risk. To the best of our knowledge, the mechanisms of this acceleration of atherosclerosis have not been studied to this date.

The VICKI study aims at furthering our knowledge on the mechanisms of atherosclerotic plaque instability by means of a prospective single-centre pilot study, by comparing:

* surrogate markers of clinical vasculo-toxicity with arterial Doppler (flow mediated reserve) as defined by the International Cardio-Oncology Society;
* circulating biomarkers

Before and after receiving ICIs for solid cancer treatment.

DETAILED DESCRIPTION:
Context. Immune checkpoint inhibitors (ICIs) are largely prescribed in a growing number of cancer diseases and at earlier stages (non metastatic cancer). Among immune-related adverse events, (iRAEs), the incidence of major cardiovascular events due to atherosclerosis reaches 13% at one year in patients at high risk. To the best of our knowledge, the mechanisms of this acceleration of atherosclerosis have not been studied to this date.

Endothelial dysfunction is a predictor of the development of atherosclerotic plaque and events related to erosion or rupture. Endothelial dysfunction correlates well with the increase of circulating microparticles in various populations. The increase of circulating microparticles is also associated with major cardiovascular events.

The International society of Cardio-Oncology (IC-OS) recently published a definition for subclinical vascular toxicities due to ICIs. It includes non-invasive imaging methods readily available at the bedside (Herrmann et al. European Heart Journal 2022), largely replicated in the recent European Society of Cardiology (ESC) guidelines 2022. It includes the decrease of flow mediated reserve <7% or hyperhemia index <2; or the decrease of any of these biomarkers > 50% from baseline.

Aims and Methods. The VICKI study aims at furthering our knowledge on the mechanisms of atherosclerotic plaque instability by means of a prospective single-centre pilot study, by comparing:

* surrogate markers of clinical vasculo-toxicity with arterial Doppler (flow mediated reserve, hyperhemia index, plaque volume) as defined by IC-OS;
* circulating microparticles; Before and after receiving ICIs for solid cancer treatment.

The number of participants:

* 40 patients receiving ICIs for solid cancer (alone or in combination of other cancer drugs);
* 40 controls (matched by age, gender, cancer type) not treated by ICIs.

Duration of participation: up to 6 weeks. Inclusion period: 12 months.

Perspectives. The VICKI study may improve our understanding of the mechanisms of atherosclerosis mediated major cardiovascular events. If circulating biomarkers correlate well with Doppler surrogate markers of vascular toxicity, larger studies to refine prediction models could be undertaken. This would be a step forward personalized care for the prediction of major cardiovascular events on ICIs.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for first ICI therapy at our institution;
* Matched controls with cancer and no ICI therapy;

Exclusion Criteria:

* Major cardiovascular event in the past 6 months;
* Unable to provide informed consent;
* History of ICI therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Endothelial dysfunction | 6 weeks
  Surrogate marker of endothelial dysfunction : Signifiant FMD variation on ICIs as defined by the International Cardio-Oncology Society

SECONDARY OUTCOMES:
Correlation of blood biomarkers to endothelial dysfunction (surrogate marker: Flow Mediated Dilatation variation) | 6 weeks
  Increase in microparticles (CD144+, CD31+/41-, CD62e+, CD235a+, CD41+, CD11+, CD3+); cytokines (e.g., IL-1b, IFNg, TNFa, VEGF-A, C, D, HGF); single-cell profiling and deep immunophenotyping.
Major cardiovascular event (MACE) | 6 months
  Collection of clinically relevant MACE at clinical follow-up: acute coronary syndrome; coronary angioplasty; stroke; cardiac suddent death, myocarditis, myositis.

CONTACTS AND LOCATIONS:
Locations (1):
- INstitut Mutualiste Montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: No